CLINICAL TRIAL: NCT01277198
Title: The Role of Flexible Cystoscopy in Laparoscopic Stone Surgery: a Single Surgeon Experience
Brief Title: Role of Flexible Cystoscopy in Laparoscopic Stone Surgery
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Seoul National University Boramae Hospital, Seoul National University Boramae Hospital
Other Study IDs: lapastone; flexible cysto in laparo
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: Kidney Calculi; Ureteral Calculi
Keywords: kidney calculi; ureteral calculi; cystoscopes; laparoscopes
MeSH Terms: conditions — Kidney Calculi; Ureteral Calculi

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- surgery without using a flexible cystoscopy: surgery without using a flexible cystoscopy: patients who did not undergo a flexible cystoscopy during laparoscopic stone surgery
- surgery with using a flexible cystoscopy: surgery with using a flexible cystoscopy: patients who underwent a flexible cystoscopy during laparoscopic stone surgery

SUMMARY:
Authors want to investigate the usefulness of flexible cystoscopy in performing laparoscopic pyelolithotomies and ureterolithotomies by comparing operative results of a single surgeon's experience.

DETAILED DESCRIPTION:
Previous trials to increase stone clearance rates have been recently reached using flexible equipment in laparoscopic surgery, however, it is not clear whether using flexible equipment is really helpful in performing pyelolithotomies and the clearance rates using flexible equipment varies 71% to 100%. Therefore, authors plan to investigate the usefulness of flexible cystoscopy in performing laparoscopic pyelolithotomies and ureterolithotomies by comparing operative results of a single surgeon's experience.

ELIGIBILITY:
Inclusion Criteria:

* patients with complex renal stones and large or impacted ureter stones
* patients who underwent laparoscopic pyelolithotomies with concomitant calyceal stone removal or ureterolithotomy using a flexible cystoscopy or not

Exclusion Criteria:

* active infection, uncontrolled bleeding tendency, previous abdominal surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 71 patients with complex renal stones and large or impacted ureter stones. All the patients underwent laparoscopic pyelolithotomies with concomitant calyceal stone removal or ureterolithotomy using a flexible cystoscopy or not.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2005-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
the presence of residual stones | intravenous pyelogram at 12 weeks postoperatively
  We judged the success when there is no residual stone in the intravenous pyelogram at 12 weeks postoperatively

SECONDARY OUTCOMES:
stone numbers and sizes, surgical approach, insertion of a DJ ureteral catheter, and use of a flexible cystoscopy, etc | Retrospective review of data
  Preoperative evaluation included a complete history, physical examination, and imaging work-up such as X-ray or computed tomography (CT). Mean preoperative stone numbers and sizes were evaluated and we also evaluated operative information such as surgical approach, insertion of a DJ ureteral catheter, and use of a flexible cystoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Cho, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Boramae Hospital, Seoul, Seoul, South Korea